CLINICAL TRIAL: NCT03924752
Title: Development of a Powered Exoskeleton Device for Lower Limb Assistance
Brief Title: Powered Hip Exoskeleton Assistance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H19178
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Lower Limb Injury
Keywords: Exoskeleton
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Intervention Model Description: The model used is a repeated measures single arm study. Multiple conditions including using and not using the device will be tested on the same subjects to have multiple test points on a per subject basis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy individuals using powered exoskeleton (Experimental): This study will be conducted on a sample population of able-bodied subjects (single arm). Each subject will test with each condition of the exoskeleton (repeated measures).
  Interventions: Device: Powered hip exoskeleton

INTERVENTIONS:
Device: Powered hip exoskeleton — The study team will test a powered hip exoskeleton and its capability to improve locomotion.

SUMMARY:
The increased metabolic and biomechanical demands of ambulation limit community mobility in persons with lower limb disability due to neurological damage. There is a critical need for improving the locomotion capabilities of individuals who have walking impairments due to disease to increase their community mobility, independence, and health. Robotic exoskeletons have the potential to assist these individuals by increasing community mobility to improve quality of life. While these devices have incredible potential, current technology does not support dynamic movements common with locomotion such as transitioning between different gaits and supporting a wide variety of walking speeds. One significant challenge in achieving community ambulation with exoskeletons is providing an adaptive control system to accomplish a wide variety of locomotor tasks. Many exoskeletons today are developed without a detailed understanding of the effect of the device on the human musculoskeletal system. This research is interested in studying the question of how the control system affects human biomechanics including kinematic, kinetics and muscle activation patterns. By optimizing exoskeleton controllers based on human biomechanics and adapting control based on task, the biggest benefit to patient populations will be achieved to help advance the state-of-the-art with assistive hip exoskeletons.

DETAILED DESCRIPTION:
One significant challenge in achieving community ambulation with exoskeletons is providing an adaptive control system to accomplish a wide variety of locomotor tasks. Many exoskeletons today are developed without a detailed understanding of the effect of the device on the human musculoskeletal system. The study is interested in exploring the question of how the control system affects human biomechanics including kinematic, kinetics and muscle activation patterns. By optimizing exoskeleton controllers based on human biomechanics and adapting control based on task, this work will be able to provide the biggest benefit to patients and advance the state-of-the-art with assistive hip exoskeletons. A large patient population that could benefit from lower limb assistive technology are stroke survivors, which is the specific population this proposal targets. One common characteristic of stroke survivors who regain their ability to walk is that the hip muscles are overtaxed due to distal weakness. The investigators propose to use a powered hip exoskeleton to augment their proximal musculature, which needs to produce significant power output in most locomotion activities such as standing up, walking, and going up stairs or slopes. Another biomechanical aspect of stroke survivors is an asymmetric gait in terms of kinematics, kinetics and muscle activations. The research team will examine what kind of exoskeleton assistance is most beneficial to stroke survivors for enhancing community ambulation. The hypothesis is that since the gait is asymmetric, the controller will need to be asymmetric to provide optimal assistance to aid in mobility. The group's long-term research goal is to create powered assistive exoskeletons devices that are of great value to individuals with serious lower limb disabilities by improving clinical outcomes such as walking speed and community ambulation ability. The overall objective of the proposed project is to study the biomechanical effects of using a hip exoskeleton with adaptive controllers for assisting stroke survivors with lower limb deficits to improve their community ambulation capabilities. The central hypothesis overarching both aims is that exoskeleton control that adapts to environmental terrain will improve mobility metrics for human exoskeleton users on community ambulation tasks. The rationale is that since human biomechanics change based on task, exoskeleton controllers likewise need to optimize their assistance levels to match what the human is doing. The first aim of the proposed study is to determine the benefit of exoskeleton control that adapts to the environment for improving community ambulation capability. The team has previously designed and extensively tested an autonomous hip exoskeleton in able-bodied subjects on a treadmill. The investigators plan to extend their control framework to over ground walking and tune assistance magnitude and timing levels to enable efficient locomotion over stairs and ramps on their novel terrain park. The investigators plan to compare a controller that adapts its assistance strategy based on locomotion task to a static controller as well as not wearing the exoskeleton. The primary hypothesis for this aim is that exoskeleton control that adapts to environmental terrain will improve mobility metrics such as task completion speed for human exoskeleton users on community ambulation tasks. The expected outcome of these aims will be an increased understanding of the biomechanical and clinical effects in applying hip assistance with a robotic exoskeleton in community ambulation tasks such as overground walking, ramps and stairs. This work will serve as a foundational start for a broader planned study of optimizing controllers to improve biomechanics in the walking impaired using powered hip autonomous exoskeletons.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-85 years of age
* Subjects should be capable of walking, ascending/descending stairs and ramps with full capability in lower extremity passive range of motion (knee flexion contracture of >10 degrees, knee flexion ROM < 90 degrees, hip flexion contracture < 25 degrees, and ankle plantar flexion contracture of >15 degrees).
* Subjects must be able to walk for at least 5 minutes and willing and able to participate over a 1-6 hours experiment with breaks and rest enforced regularly and as needed.
* Subjects must be able to transfer (sit-to-stand and stand-to-sit) with no external support (arm rests OK) and to ambulate over small slopes (3 degrees) and a few steps (6 steps).

Exclusion Criteria:

* History of neurological injury, gait pathology, or cardiovascular condition that would limit your ability to ambulate for multiple hours.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-13 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Young, Ph.D., Principal Investigator — Georgia Tech
Locations (1):
- Exoskeleton and Prosthetic Intelligent Controls Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy and young individuals were recruited between February 2021 to March 2021. The first participant was enrolled on February 2021 and the last participant was enrolled on March 2021.
Groups:
- Healthy Individuals Using a Powered Hip Exoskeleton: This study will be conducted on a sample population of able-bodied subjects (single arm). Each subject was tested with each condition of the exoskeleton (repeated measures).
  Powered hip exoskeleton: The study team tested a powered hip exoskeleton and its capability to improve locomotion.
Period: Overall Study
Arm/Group | Healthy Individuals Using a Powered Hip Exoskeleton
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Individuals Using a Powered Hip Exoskeleton
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Height [Mean (Standard Deviation); unit: centimeters] | 174.06 (6.35)
weight [Mean (Standard Deviation); unit: kilograms] | 69.8 (8.1)
Self-Selected Walking Speed [Mean (Standard Deviation); unit: meters per second] — The subject's baseline preferred walking speed in the different walking conditions was recorded. Five walking conditions were evaluated: 1) level-ground, 2) ramp ascent, 3) ramp descent, 4) stair ascent and 5) stair descent. The ramp incline was set to 9.2 degrees and the stair height was set to 15.24 cm. The walking speed was calculated by looking at the distance traveled divided by time. The distance was fixed and a completion time for each trial was recorded with a computer timer to calculate the average walking velocity for a given trial.
  meters per second
    Level-Ground | 1.08 (0.14)
    Ramp Ascent | 1.31 (0.06)
    Ramp Descent | 1.27 (0.17)
    Stair Ascent | 0.62 (0.07)
    Stair Descent | 0.69 (0.06)

OUTCOME MEASURES:

1. Primary Outcome: Self-Selected Walking Speed Using Hip Exoskeleton Assistance Across Different Locomotion Modes
Description: Measure Description: The subject's preferred overground walking speed while wearing a powered hip exoskeleton was recorded. During walking, the exoskeleton provided hip assistance. There was a total of five walking conditions that were evaluated: 1) level-ground, 2) ramp ascent, 3) ramp descent, 4) stair ascent and 5) stair descent. The ramp incline was set to 9.2 degrees and the stair height was set to 15.24 cm. The user's preferred walking speed was calculated by looking at the distance traveled divided by time for a given walking condition. The distance was fixed and a completion time for each trial was recorded with a computer timer to calculate the average walking velocity for a given trial.
Time Frame: 4 hours
Population: The effect of hip exoskeleton assistance on the subject's preferred overground walking speed across different locomotion modes was evaluated. Five walking conditions were 1) level-ground, 2) ramp ascent, 3) ramp descent, 4) stair ascent, and 5) stair descent. The ramp incline was set to 9.2 degrees and stair height was set to15.24 cm. During walking, the exoskeleton provided assistance relevant to the user's biological demand (hip flexion and extension assistance).
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Healthy Individuals Using a Powered Hip Exoskeleton
Number analyzed (Participants) | 10
meters per second
  Level-Ground Assistance | 1.14 (0.08)
  Ramp Ascent Assistance | 1.26 (0.08)
  Ramp Descent Assistance | 1.26 (0.15)
  Stair Ascent Assistance | 0.61 (0.05)
  Stair Descent Assistance | 0.71 (0.07)
Statistical Analysis 1: Comparison: Healthy Individuals Using a Powered Hip Exoskeleton; Test type: Other — A two-way repeated-measures analysis of variance (ANOVA) was performed on different walking conditions (including the baseline of not wearing the exoskeleton) on the subject's overground self-selected walking speed across different locomotion modes by setting the significant value to 0.05. Two independent variables were assistance type (Exo vs No Exo) and different locomotion modes; p = 0.9547, ANOVA — This presents the effect of exoskeleton assistance on the user's preferred overground walking speed across different locomotion modes

ADVERSE EVENTS:
Time Frame: Duration of the experiment (4 hours)
Description: The total number at risk for serious adverse events is 10 (number of participants). The main event that we would consider a serious event is if the subject falls during the trial when the exoskeleton is providing assistance. We monitored this serious event throughout the data collection but did not observe any.
Arm/Group | Healthy Individuals Using a Powered Hip Exoskeleton
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT03924752/Prot_003.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT03924752/SAP_002.pdf
  • Informed Consent Form (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT03924752/ICF_000.pdf